CLINICAL TRIAL: NCT04402502
Title: Dynamic 4DCT to Examine the Effect of Mal-united Distal Radius Fractures on Carpal Contact Mechanics
Brief Title: Dynamic 4DCT to Examine Wrist Carpal Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5147
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis
Keywords: 3D Ultrasound Monitoring
MeSH Terms: conditions — Osteoarthritis | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Healthy Population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Population (Experimental): Healthy Individuals with no presence of neurological disorders, rheumatoid arthritis or comorbid health conditions, and are not pregnant.
  Interventions: Device: Ultrasound Imaging

INTERVENTIONS:
Device: Ultrasound Imaging — The participant will go to the Rheumatology clinic (St. Joseph's Hospital) and have 3D hand ultrasound performed on their hands.

SUMMARY:
Osteoarthritis can develop after an injury like a broken bone. Problems with how the bones line up can lead to abnormal loading which will destroy the cartilage that covers and protects the bones. Once this happens, patients experience substantial pain and disability. Researchers and doctors use planar x-rays to evaluate joints; but these are not always precise and are limited to two dimensions. Three-dimensional (3D) computed tomography (CT) can be used to look at the joints of the wrist in three dimensions, but is limited to static frames. Symptoms arising from joint instability often occur when the wrist is moving and when it is performing a functional task (opening a jar). Four dimensional computed tomography (4DCT) can detect dynamics changes in the small structures of the wrist with high temporal and spatial resolution. This novel imaging techniques provides a movie of bones in the wrist, in 3D, while in the scanner. In this proposal, the investigator's will use 4DCT and look at how joint alignment of the distal radius effects the joints in the wrist, and investigate how it relates to patient's function, description of pain and the presence of Osteoarthritis 10 years following fracture. This imaging will drive safer clinical research and practice and will develop tools that predict the risk of developing arthritis that will help doctors determine when surgery is necessary to prevent arthritis of the hand and wrist, and pain and disability.

DETAILED DESCRIPTION:
A series of 60 participants (30 male: 30 female) with current distal radius fractures will be recruited. Clinical eligibility will include a unilateral DRF treated with closed reduction and casting. These measures will be assessed at baseline (<6 weeks following injury), 3- 6 months and 12 months following fracture. A second series of 80 participants (40 male: 40 female) who suffered a DRF ≥10 years previously will be recruited and tested. Exclusion criteria for these two cohorts will include presence of neurological disorders, rheumatoid arthritis or co-morbid health conditions that preclude completion of study measures. Twenty additional healthy participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English, capacity to provide consent,
* over the age of 18 years old, with no previous injury to either hand or wrist

Exclusion Criteria:

* pregnancy and presence of neurological disorders, rheumatoid arthritis or comorbid health conditions that preclude completion of study measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Hand Joint Spacing | 3 years
  To measure joint spacing of the hand in a 3D ultrasound image

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada